CLINICAL TRIAL: NCT00504972
Title: Phase I Trial of Anti-CD74 (hLL1) Antibody Therapy in B Cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0608008669
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — milatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Treatment (Experimental): This study is a single arm study
  Interventions: Drug: hLL1

INTERVENTIONS:
Drug: hLL1 — hLL1 administered intravenously once daily Monday through Friday for 2 consecutive weeks (10 total doses) at one of 4 planned dose levels: 1.5, 4, 6 or 8 mg/kg.

SUMMARY:
Previous experience with antibody therapy in both NHL and CLL warrants further exploration of new antibody treatments for these diseases.

Immunomedics has developed hLL1 (previously designated EPB-1), which is a CDR-grafted, fully humanized monoclonal antibody specifically targeting CD74.38 The human IgG1 backbone for hLL1 is the same as hLL2 (epratuzumab), a monoclonal antibody whose safety has been demonstrated in clinical trials of patients with B-cell malignancies and autoimmune disorders.

This is a Phase I, open-label, study conducted in patients with recurrent non-Hodgkin's lymphoma (NHL) or chronic lymphocytic leukemia (CLL) who have progressed after at least one prior standard treatment. All patients will receive hLL1 administered intravenously once daily Monday through Friday of each of 2 consecutive weeks (10 total doses.) Patients will be assigned to a cohort for hLL1 treatment dose assignment (escalating doses of hLL1 per statistical plan) in order to determine the maximum tolerated dose (MTD) for this administration schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of recurrent B cell non-Hodgkin's lymphoma or diagnosis of recurrent chronic lymphocytic leukemia
* Patient has received at least one prior treatment with standard chemotherapy and at least one prior treatment with rituximab (negative HAHA test required if received prior humanized antibody treatment)
* Patient has not received anti-cancer therapy within 28 days of treatment unless disease progression has been demonstrated and toxicities from prior therapy have resolved
* Available tumor tissue (lymph node/mass, blood or bone marrow) for correlative analyses (paraffin or frozen, recent or archived)
* Measurable disease as defined by a tumor mass > 1.5 cm in one dimension or WBC > 5,000 (CLL patients)
* Age > 18 years
* Patient has KPS > 50%
* Absolute granulocyte count > 1000 cells/mm3
* Platelet count > 50,000 cells/mm3
* Creatinine < 2.0 x ULN
* Total bilirubin < 2.0 x ULN
* Patient agrees to use birth control if of reproductive potential
* Patient has signed IRB-approved informed consent

Exclusion Criteria:

* Known central nervous system (CNS) involvement by lymphoma
* Known HIV disease
* Patient is pregnant or nursing
* Patient is receiving other investigational drugs
* Known serum human anti-human antibodies (HAHA)
* Estimated life expectancy of < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-06; Primary Completion 2011-04-01 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
To determine the toxicity profile and maximum tolerated dose (MTD) of hLL1 when administered to patients with recurrent non-Hodgkin's lymphoma and chronic lymphocytic leukemia | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: John P Leonard, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided